CLINICAL TRIAL: NCT03537040
Title: A Pilot Study to Assess the Feasibility and Acceptability of a Novel Intervention to Help People Think About Their Neuroleptic Medication Use.
Brief Title: Piloting MOL Intervention for Neuroleptic Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Rea Dicks, Trainee Clinical Psychologist, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 238098
Record Dates: First submitted 2018-04-18; First posted 2018-05-25 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Psychosis; Medication Adherence
MeSH Terms: conditions — Psychotic Disorders; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Method of Levels (Other): Talking therapy- duration and frequency of sessions to be determined by participant
  Interventions: Other: Method of Levels

INTERVENTIONS:
Other: Method of Levels — Talking Therapy

SUMMARY:
The aim of the current study is to pilot a novel intervention to help people explore their decision making around the use of neuroleptic medication. A case series design will be used, with outcome variables measured at multiple time points pre-, during- and post-intervention. Participants will also be asked to complete an evaluation interview post-intervention. The primary aim is to investigate the feasibility and acceptability of offering the intervention.

DETAILED DESCRIPTION:
Many service users experiencing psychosis are prescribed neuroleptic medication as the core component of treatment. However, discontinuations rates are high, which may be influenced by poor response rates and scepticism about the value of medication.

Frequently people discontinue without professional involvement, which is associated with negative outcomes. It is a particularly high risk period for relapse, especially if withdrawal is done quickly. There is an urgent need to advance practices in helping service-users to make a decision regarding neuroleptic medication that can then be supported by clinicians.

Current interventions regarding medication use predominantly focus on increasing adherence to medication regimes using, for example, financial incentives. This raises ethical concerns over the potential for service users' priorities and preferences to be disregarded, leading to increased coercion and reduced empowerment for service users. The recovery movement emphasises the need to understand personal priorities when considering treatment options and informed choice and shared-decision making is promoted by government initiatives and practice guidelines.

Shared decision-making commonly occurs within physical health settings. Patient decision aids have been found to improve patients' knowledge of available options and help patients to have more accurate expectations of potential benefits and harms, reach choices that are more consistent with personal values and participate in decision making. Despite this, shared-decision making has not been adopted more widely and is particularly poor within mental health settings.

The current study aims to explore the feasibility and acceptability of an intervention aimed at helping service users in mental health services think about their own personal priorities and decision-making around medication use. Current psychological interventions, such as cognitive behavioural therapy (CBT) and motivational interviewing (MI), view decision-making in terms of individuals making cost-benefit analyses, which then informs their "planned" behaviour. Such interventions thus target the identification of desirable medication related behaviours and then help the individual to make those behaviours occur.

Perceptual Control Theory (PCT) offers an alternative framework in which to understand medication related decision-making and behaviour. PCT regards all behaviour as goal directed but states that individuals control their experiences (or input) not their behaviour (or output). From this perspective, behaviour is understood as a means by which an individual resolves discrepancies between how they currently experience something (a current perception) and the way they want that experience to be. There is recognition that people are usually unaware of many of the different priorities (or goals) they hold, although these priorities/ goals are often incompatible (in conflict). An intervention informed by PCT (Method of Levels; MOL) would, therefore, target increasing an individual's awareness of the different personal priorities/ goals they hold in relation to medication use. The intervention would focus on exploring conflict between personal priorities, as from a PCT perspective; conflict is what causes ambivalence or difficulties in being able to enact certain planned behaviours. The aim in the current study would be to use MOL to help people develop their awareness of what is important to them in relation to medication use, as opposed to focusing on planning specific behaviours.

The aim in the current study would be to use MOL to help people explore their decision around the use of neuroleptic medication. Traditionally the focus of a MOL session is determined by the client and can vary from person to person, however, for this study the sessions will be specifically focused on neuroleptic medication use. The sessions will aim to help people explore a range of thoughts and feelings about decisions around medication use and how these relate to other important life values and goals. Another key aim of sessions will be to help people develop awareness of conflicts in their goals so that they might begin to find potential resolution. Due to the nature of the intervention being very patient-led and idiosyncratic, the outcome will vary from person to person. The intervention does not attempt to increase adherence or encourage discontinuation to the neuroleptic medication. It aims to help people develop awareness of how they feel about using neuroleptic medication and how medication might relate to other things that are important to them in life.

If this is a feasible and acceptable approach to use then future research would explore whether prescribers could incorporate this approach to working in their consultations with service users.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years of age
* Capacity to provide informed written consent
* Able to converse in English proficiently
* Currently under the care of an Early Intervention Service or Community Mental Health Team
* Ambivalent around medication use
* Experience of psychosis
* Be able to be assessed in an outpatient facility (exceptions will be made for disabilities)

Exclusion Criteria:

* If currently experiencing such a deterioration in mental state that they may have difficulties making decisions in their life
* If significant risk of harm to self or others is present
* If there is an organic basis for psychosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited to the study | through study completion, an average of 5 months.
  Number of participants recruited to the study
Number of participants retained during the study | through study completion, an average of 5 months.
  Number of participants retained during the study
Change in therapeutic alliance from baseline to 12 weeks | baseline, 12 weeks.
  The Session Rating Scale is a brief therapeutic alliance measure designed for every session clinical use. The SRS is a four-item visual analogue instrument that explores the relationship, goals and topics, approach or method, and how the client perceives the session in total. Scores range between 0 and 40, higher scores suggest better therapeutic alliance.

SECONDARY OUTCOMES:
Change in treatment-related empowerment from baseline to 12 weeks | baseline, 12 weeks.
  The Treatment-related Empowerment Scale assesses the patients perceived degree of involvement within their treatment by assessing components of communication, treatment choice, decisions and satisfaction. The scale consists of 10 items in which respondents rate the extent to which their experience matches each statement on a 5 point Likert scale. High scores represent higher treatment-related empowerment.
Change in attitude towards medication from baseline to 12 weeks | baseline, 12 weeks.
  The Drug Attitude Inventory-10 a 10-item modified version of the Drug Attitude Inventory-30 Questionnaire, commonly used to evaluate medication adherence and captures an individual's general attitude about taking medication. Scores range between -10 and +10, higher scores indicate a more positive attitude towards medication.
Change in compliance to medication regime from baseline to 12 weeks | baseline, 12 weeks.
  Participants will be asked to rate their current compliance using a 4-point scale that was developed for another study (Barrowclough et al., 1999). Scores range from 0-4, higher scores indicate higher compliance.
Change in personal recovery from baseline to 12 weeks | baseline, 12 weeks.
  Questionnaire about the Process of Recovery a 15-item measure used to assess personal recovery. Scores range between 15 and 75, higher scores are indicative of recovery.
Change in engagement with services from baseline to 12 weeks | baseline, 12 weeks.
  The Service Engagement Scale is a 14-item clinician-rated measure that assesses service user engagement with community mental health services. Scores range between 0 and 42, lower scores indicate better engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tai, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - Lancashire Care NHS Foundation Trust, Preston, Lancashire
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Annoymous data files for outcome data will be shared on request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by research team. Requestors will be required to sign a data access agreement

REFERENCES:
- [Background] Moncrieff J. Does antipsychotic withdrawal provoke psychosis? Review of the literature on rapid onset psychosis (supersensitivity psychosis) and withdrawal-related relapse. Acta Psychiatr Scand. 2006 Jul;114(1):3-13. doi: 10.1111/j.1600-0447.2006.00787.x. PMID 16774655
- [Background] Mansell W, Carey TA. A century of psychology and psychotherapy: is an understanding of 'control' the missing link between theory, research, and practice? Psychol Psychother. 2009 Sep;82(Pt 3):337-53. doi: 10.1348/147608309X432526. Epub 2009 Apr 1. PMID 19341533